CLINICAL TRIAL: NCT06889337
Title: A Comparative Study of Supine Position and the Head Elevated Position on the Level of Sensory Block After Spinal Anesthesia in Morbidly Obese Parturient Undergoing Elective Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MRC-01-21-032
Record Dates: First submitted 2025-02-23; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: High BMI

STUDY DESIGN:
Intervention Model Description: Total 90 patients will be enrolled in the study, 45 patients in each group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEAD ELEVATING LARYNGOSCOPY PILLOW (Experimental): the head elevation beyond the sniffing position, also known as ramped position or head elevated laryngoscopy position, usually achieved by specially designed pillows such as the Oxford head elevating laryngoscopy pillow (Alma Medical, Oxford, UK) or the Troop® elevation pillow (Mercury Medical, Clearwater, FL, USA)
  Interventions: Other: head elevated laryngoscopy position by Oxford pillow
- Standard pillow group (No Intervention): Standard pillow group

INTERVENTIONS:
Other: head elevated laryngoscopy position by Oxford pillow — ramped position, also known as head elevated laryngoscopy position,
  Arms: HEAD ELEVATING LARYNGOSCOPY PILLOW

SUMMARY:
The sniffing position defined as neck flexion with upper cervical extension, is traditionally recommended for general anesthesia induction, as it improves laryngoscopic views. However, the head elevation beyond the sniffing position, also known as ramped position or head elevated laryngoscopy position, usually achieved by specially designed pillows such as the Oxford head elevating laryngoscopy pillow (Alma Medical,Oxford, UK) or the Troop® elevation pillow (Mercury Medical, Clearwater, FL, USA)has been shown to not only increase respiratory reserve but also to improve laryngeal views in patients undergoing bariatric surgery. Additionally it helps in pre-oxygenating the patient more efficiently by keeping the airway patent and provides easier bag-mask ventilation.

It may also benefit the term parturient in a similar way by improving functional residual capacity (FRC), ventilation and comfort. However, this positon may affect the cephalad spread of the intrathecal local anesthetic.

Two earlier studies looked at the intrathecal local anesthetic spread in obstetric patients when placed in the head elevated laryngoscopy position, and both suggested poor cephalad spread, with patients requiring higher supplementation.

However, both studies excluded morbidly obese patients. The Investigators hypothesized that in obese parturients with BMI more than or equal 40, higher intra-abdominal pressures and possibly lower CSF volumes will counteract the poor cephalad spread associated with this position. The aim of this study is to determine the effect of a ramped position on intrathecal local anesthetic spread in the morbidly obese term parturients with BMI more than or equal 40 undergoing elective Cesarean delivery(CD).

ELIGIBILITY:
Inclusion Criteria:

* Age 18yrs of age or more
* BMI 40 or more and more than or equal 37 weeks of gestation
* elective CD
* consented for neuraxial anesthesia
* singleton fetus
* ASA class 3 (no co-morbidities except morbid obesity, gestational diabetes, and gestational hypothyroidism)

Exclusion Criteria:

* Age <18 years
* BMI less than 39.9 and <37 weeks of gestation
* parturient preference for general anesthesia or contraindication to neuraxial anesthesia
* Women with comorbidities other than obesity, gestational diabetes or gestational hypothyroidism.
* women in active labor (>3 cm dilated with regular uterine contractions)
* emergency CD
* Possible uterine over-distension or under-distension (e.g. polyhydramnios, estimated fetal weight >4 kg by ultrasound scan, or oligohydramnios or concern for fetal IUGR)
* maternal height <150 cm or >180 cm.
* Patients for which more than 2 minutes is taken in positioning after anesthesia induction (Time 0).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 90 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
The sensory level (loss of cold and pin prick sensation) at 15 min after the intrathecal administration of the medication in the parturient | From date of randomization until the date of first documented progression, assessed up to 48 months

SECONDARY OUTCOMES:
Incidence of inadequate block level at 15 min and need for epidural supplements | From date of randomization until the date of first documented progression, assessed up to 48 months
  Secondary Outcomes:
  I. Incidence of inadequate block level at 15 min II. The need for epidural supplementation. III. Dosage of epidural local anesthetics to achieve adequate block level following the spinal anesthetic.
  IV. The need and dosage of iv opioids for intraoperative supplemental analgesia V. The incidence of pain throughout the procedure (by the use of NRS). VI. The use and dosage of vasopressor. VII. The rate of conversion to general anesthesia. VIII. Maternal satisfaction with the position. IX. Neonatal outcomes (Birth weight in kilograms, APGAR scores, umbilical cord gases and lactate)

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar